CLINICAL TRIAL: NCT07274202
Title: The Physical and Mental Impact of ART: an RCT Comparing IVM and Conventional Ovarian Stimulation From a Patient Perspective
Brief Title: The Physical and Mental Impact of ART: IVM vs Conventional Ovarian Stimulation
Acronym: QolART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BUN1432025000250
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
Keywords: physical side effects; mental side effects; In vitro maturation; conventional ovarian stimulation
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVM (Experimental): treatment with in vitro maturation
  Interventions: Other: Questionnaires
- cOS (Active Comparator): treatment with conventional ovarian stimulation
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Three types of questionnaires will be completed: FERTIQoL, HADS en self-developed questionnaire for side-effects of treatment type. Qoestionnaires will be completed at 7 different timepoints

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is one of the most common endocrine conditions, affecting around 10% of women in reproductive age (ESHRE PCOS guideline, 2023).

PCOS is a heterogeneous condition characterized by a combination of Polycystic Ovarian Morphology (PCOM) on ultrasound scan, oligo- or amenorrhea and/or hyperandrogenism. Women diagnosed with PCOS are known to have a higher risk for type 2 diabetes mellitus, cardiovascular pathology, pregnancy complications and an impaired quality of life (QoL) (Borghi et al., 2017; ESHRE guideline, 2023). Conventional Ovarian Stimulation (cOS) followed by in vitro fertilization (IVF) or intra cytoplasmic sperm injection (ICSI) is the most frequently used type of ART for PCOS patients. However, women with PCOS often exhibit ovarian hyperresponse to conventional-dose gonadotropin stimulation/cOS, with ovarian hyperstimulation syndrome (OHSS) as the most frequently occurring iatrogenic complication (Vesztergom et al., 2021 ; ESHRE PCOS guideline, 2023). Although, due to a number of strategies to prevent OHSS, the occurrence of severe OHSS has almost been eliminated, with the use of GnRH agonists for final oocyte maturation instead of an hCG trigger as the most efficient strategy, patients might still experience symptoms of abdominal pain and bloating as an indication for mild or moderate OHSS (Bodri et al., 2010 ; Shrem et al., 2019). Aside from the risk for OHSS, patients undergoing cOS, which represents on average a two-week hormonal treatment, may also experience symptoms of hot flushes, breast tenderness, mood swings and higher psychological burden resulting in a reduced QoL during fertility treatment (Barrière et al., 2019; Shrem et al., 2019 ; Adeleye et al., 2020).

In view of the aforementioned inconveniences of cOS, In Vitro Maturation of oocytes (IVM) followed by ICSI has been proposed as an alternative treatment option in a PCOS population (Trounson et al., 1994 ; ESHRE PCOS guideline, 2023). In Vitro Maturation has been labeled as a more 'patient-friendly' approach, with the ability to further eliminate the risk for OHSS, minimize cycle monitoring (resulting in less in-hospital visits) and reduced side-effects from hormonal ovarian stimulation (Gilchrist and Smitz, 2023; ESHRE PCOS guideline, 2023 ; Vuong et al., 2023). However, to the best of our knowledge, there is only limited research that investigated the prevalence and types of side-effects and the impact on pain scores and QoL of IVM treatment in PCOS patients (Sanmartin et al., under review; Marchante et al., 2024). Therefore, we set out to investigate the impact of IVM on pain scores, side-effects and QoL during fertility treatment in women diagnosed with severe PCOS. We defined severe PCOS as women with a serum AMH>10ng/mL because we observed that above this cut-off, cumulative ongoing pregnancy rates were non-inferior after IVM compared to cOS (Mostinckx et al., 2024), with non-inferiority defined as a difference of less than 10% in cumulative ongoing pregnancy rate per cycle.

This trial is a single center, superiority, randomized controlled trial that will be conducted at Brussels IVF, UZ Brussel, Belgium in a PCOS population, presenting for their first round of ART at Brussels IVF. Each patient can only participate once in this trial.

64 patients are planned to be enrolled in the trial. 32 patients will be required in the control group (cOS group) and 32 patients in the interventional group (IVM group).

Patients will randomly undergo IVM or cOS following randomization. Both treatments will be executed as per treatment as usual (TAU). In both treatment arms, included patients and their partners, will be asked to complete questionnaires at different timepoints after randomization into one of the two treatment arms:

* At the time of counseling (T1)
* At the end of stimulation (T2)
* On the day of oocyte retrieval (T3)
* On the day after oocyte retrieval (T4)
* At 7 days after oocyte retrieval (T5)
* At the end of first embryo transfer cycle (T6)
* End of first ART cycle Used questionnaires are two validated questionnaires, FertiQoL and HADS, and a questionnaire developed to investigate side-effects and pain scores after oocyte retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Age from >18 to <35 years
* Patients with a PCOS diagnosis: The PCOS diagnosis will be based on the ESHRE PCOS guideline (2023) and the evidence-based methodology workshop on polycystic ovary syn-drome, December 3-5, 2012 using the following classification: Phenotype A (hyperandro-genism + oligo-/amenorrhea + PCOM), Phenotype C (hyperandrogenism + PCOM) and Phenotype D (oligo-/amenorrhea + PCOM). Hyperandrogenism is defined as the presence of clinical and/or biochemical hyperandrogenism following the ESHRE PCOS guideline, 2023. Oligomenorrhea or amenorrhea is considered as an average cycle duration > 35 days.
* A serum AMH concentration of >10.00 ng/ml as measured using the Elecsys platform by Roche at UZ Brussel. Threshold of 10 ng/mL or higher was adopted based on the result of a multivariable analysis by our group (Mostinckx et al. (2024)), which showed that ongoing pregnancy rates in women with AMH of 10ng/mL or higher did not depend on the type of treatment (IVM vs. cOS).
* Embarking on their first round of ART treatment at Brussels IVF.
* Eligible for ART either because previous treatment with ovulation induction failed and/or because of male factor infertility.
* Patients must be able to speak Dutch, French or English.

Exclusion Criteria:

* BMI <18 or >35 kg/m²
* Patients with a general anesthesia during oocyte retrieval
* Patients with a PCOS phenotype B will be excluded from the trial since these patients do not polycystic ovaries on ultrasound scan and are therefore not considered hyperrespond-ers.
* Patients who do not have a partner
* Need for preimplantation genetic testing (PGT)
* high grade endometriosis (> grade 2)
* Couples who need donor oocytes

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Pain after oocyte retrieval | From enrollment to the end of treatment or one year after radnomization